CLINICAL TRIAL: NCT05013853
Title: Clinical Performance Resin Bulk Fill Dual-cured of Posterior Restorations: Clinical Study
Brief Title: Resin Bulkfill Dual-Cured of Proximal Restoration. Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Patricio Vildosola Grez, Clinical Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROPRGFO_002019.25.
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Dental Restoration; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resin Z350 of proximal posterior teeth (Active Comparator): Restorative with Z350 composite of proximal caries lesions or restorations replacement
  Interventions: Procedure: Restoration teeth
- Resin Tetric N Ceram Bulkfill of proximal posterior teeth (Active Comparator): Restorative with Tetric N Ceram Bulkfill composite of proximal caries lesions or restorations replacement
  Interventions: Procedure: Restoration teeth
- Resin Fill Up! of proximal posterior teeth (Experimental): Restorative with Fill Up! composite of proximal caries lesions or restorations replacement
  Interventions: Procedure: Restoration teeth

INTERVENTIONS:
Procedure: Restoration teeth — Remove caries and restore with resin composite

SUMMARY:
Objective: To evaluate the immediate clinical performance using FDI criteria in occlusal and proximal lesions restored with dual polymerization bulkfill composite resin.

Materials and methods: Experimental, clinical, controlled, randomized, double-blind study. For the evaluation of Fill-up! (FU) will be clinically compared to the control groups of a conventional Tetric N-Ceram (TB) RBK and Filtek z350 (z350) conventional composite resin. The adhesive process will be carried out under absolute isolation, of selective etching of 37% orthophosphoric acid enamel before applying the respective adhesive according to the trademark of the composite resins. The evaluation will be to 30 days, 6, 12, 18 and 24 months using the modified FDI criteria of postoperative sensitivity, marginal staining, color, marginal adaptation and anatomy, being 1: Excellent, 2: Good, 3: Fair, 4: unsatisfactory and 5: unacceptable. The non-parametric Kruskal Wallis test and Friedman (95% significance) used to compare the criteria.

DETAILED DESCRIPTION:
Prior to the removal of carious lesions, the tooth will be first anesthetized. The lesion areas will be prepared with a diamond rotary instrument (801G.FG.016, Jota AG Rotary Instruments - Switzerland) at high speed and under refrigeration with abundant water. Only damaged tissue conservatively removed. The corresponding measurements it recorded with a millimeter probe (Hu Friedy®, North Carolina, Chicago, USA). Prior to the insertion of the material, the sectional matrix system and the palodent type matrix system and with a wooden wedge will be used. The manufacturer's instructions for each brand of composite resin will be followed. It conditioned with 37% phosphoric acid only in enamel, wash for twice as long and dried. The corresponding adhesive will be used f Single Bond Universal adhesive (3M-Espe, ST. Paul, MN, USA) applied for the z350 group, Tetric N-Bond Universal adhesive (Ivoclar Vivadent AG, Schaan, Liechtenstein) for TB group and One Coat adhesive (Còltene, Whaladent Inc.) for FBK group. In the case of the FBK group, a final layer of Brilliant EverGlow composite resin (Còltene, Whaladent inc) will be added. Figure 3 Photopolymerization procedures performed using an LED light source with a minimum power of 1,100 mW / cm2 (Bluephase Style, Ivoclar Vivadent, AG, Schaan, Liechtenstein). The centric and eccentric occlusal contacts were verified and adjusted. For the finishing and polishing of both protocols, flexible discs (3M ESPE, St. Paul, USA) and the Enhance system (Dentsply, Petrópolis, RJ, Brazil) were used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,
* high cariogenic risk,
* availability for clinical follow-up,
* have at least 3 teeth with occlusal and / or proximal carious lesions of molars or premolars with occlusal and proximal contact,
* lesions less than 1/3 of inter-cuspal distance and depth> 3 mm in the cervical-occlusal direction and margin on enamel

Exclusion Criteria:

* Impossibility wash their teeth
* evidence of xerostomia
* uncontrolled periodontal disease,
* pregnant or breastfeeding
* bruxism or with temporomandibular disorder
* history of allergy to acrylic or its derivatives,
* portador of removable prostheses endodontically treated teeth
* cracked teeth and periapical pathology or pulp pathology symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Compare clinical performance restorations | Baseline
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI system , Unit is Ranking system has 5 scores for each different criterion. Either restoration is clinically 1: excellent, 2: good, 3:sufficient, 4: unsatisfactory, 5: clinically poor.
Compare clinical performance restorations | 6 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI system , Unit is Ranking system has 5 scores for each different criterion. Either restoration is clinically 1: excellent, 2: good, 3:sufficient, 4: unsatisfactory, 5: clinically poor.
Compare clinical performance restorations | 12 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI system , Unit is Ranking system has 5 scores for each different criterion. Either restoration is clinically 1: excellent, 2: good, 3:sufficient, 4: unsatisfactory, 5: clinically poor.
Compare clinical performance restorations | 18 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI system , Unit is Ranking system has 5 scores for each different criterion. Either restoration is clinically 1: excellent, 2: good, 3:sufficient, 4: unsatisfactory, 5: clinically poor.
Compare clinical performance restorations | 24 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI system , Unit is Ranking system has 5 scores for each different criterion. Either restoration is clinically 1: excellent, 2: good, 3:sufficient, 4: unsatisfactory, 5: clinically poor.

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Vildosola, Principal Investigator — Universidad Andre Bello
Locations (1):
- Patricio Vildosola Grez, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No